CLINICAL TRIAL: NCT03340272
Title: PROspective Multicenter Observational Study on Elective Pelvic Nodes (PRO-EPI) Irradiation in Patients With Intermediate/High/Very High Risk Prostate Cancer
Brief Title: PROspective Multicenter Observational Study on Elective Pelvic Nodes Irradiation.
Acronym: PRO-EPI
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Collaborators: Takeda (Industry)
Responsible Party: Principal Investigator, Michela Buglione, Prof, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Other Study IDs: NP2283
Record Dates: First submitted 2017-10-30; First posted 2017-11-13 (Actual); Last update posted 2020-03-18 (Actual); Status verified 2020-03

CONDITIONS: Intermediate Risk Prostate Cancer; High Risk Prostate Cancer
Keywords: prostate cancer; pelvic irradiation; hormonal treatment
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The general aim of the study is to describe the use of elective pelvic node irradiation (ENI) in Italy, in patients with intermediate/high/very high-risk prostate cancer patients submitted to adjuvant or radical Radiation Therapy (RT) with or without concomitant Androgen Deprivation hormone Therapy (ADT).

The study aims at the definition of survival, toxicity and QoL data in a representative sample of intermediate, high and very high risk prostate cancer patients consecutively recruited in Italian Radiation Oncology Center over two years.

DETAILED DESCRIPTION:
Clinical features and outcomes of the patients included in the study will be assessed as better detailed in the following lines:

1. To define the diffusion of the practice of treating pelvic lymph-nodes in patients affected by intermediate/high/very high risk non-metastatic prostate cancer (PCa) among Italian Radiation Oncology Centers, submitted to radical or post-operative radiotherapy;
2. To define the diffusion of the different radiotherapy techniques used to treat pelvic nodes and the other features of the radiation treatment;
3. To register prospectively biochemical and clinical failure, prostate cancer deaths and deaths for any cause in the population studied;
4. To register prospectively the toxicity due to radiotherapy and androgen deprivation therapy in patients treated with pelvic nodes radiotherapy;
5. To compare clinical outcomes and toxicities observed in the different clinical and therapeutic subgroups with the corresponding historical data relative to PCa patients treated with radiotherapy with or without elective pelvic nodal irradiation, already available in the existing Italian Society of Radiation Oncology databases;
6. To exploit the collected data to define the need and the features of a prospective randomized trial evaluating the efficacy of elective pelvic nodal irradiation in patients with intermediate/high/very high risk non-metastatic prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Men older than or aged 18 years;
* Histologically confirmed intermediate, high or very high risk prostate cancer patients (NCCN classification: Intermediate Risk T2b and T2c or Gleason Score 7 or Prostate specific antigen (PsA) value between 10 and 20 ng/mL; High risk: T3a or Gleason score 8-10 or PSA > 20 ng/ml; Very high risk: T3b-T4 or patients with multiple adverse risk factors reported in the high risk category that may be shifted in the very high risk group
* Patients eligible for -and actually submitted to- radical radiotherapy treatment (+/- androgen deprivation) or adjuvant radiotherapy treatment after surgery (radical prostatectomy +/- pelvic lymphadenectomy);
* No other synchronous or previous malignant tumor other than skin basal cell carcinoma;
* Patients able to understand and sign the appropriate informed consent;
* Patients able to fill the QoL questionnaire;

Exclusion Criteria:

* Patients aged less than 18;
* Patients not eligible for -and actually not submitted to- radical radiotherapy treatment (+/- androgen deprivation) or adjuvant radiotherapy treatment after surgery (radical prostatectomy +/- pelvic lymphadenectomy);
* Low risk prostate cancer (<T2b and T2c or < Gleason Score 7 or PSA value < 10 ng/mL);
* Patients with synchronous or previous malignancy other than skin basal cell carcinoma;
* Patients able to understand and sign the appropriate informed consent (IC) who decide not to subscribe IC;
* Patients not able to understand and sign the appropriate informed consent (IC)
* Patients unable to fill the QoL questionnaire.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients treated for prostate cancer without or after surgery, with or without association of hormonal treatment.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Actual)
Dates: Start 2017-02-21 (Actual); Primary Completion 2020-02-21 (Actual); Study Completion 2023-02-21 (Estimated)

PRIMARY OUTCOMES:
Practice of pelvic irradiation | Four months after the end of the enrollment
  Evaluate the number of patients treated with RT on pelvic lymph-nodes in patients affected by intermediate/high/very high risk non-metastatic prostate cancer

SECONDARY OUTCOMES:
Radiotherapy techniques used for prostate cancer irradiation | Four months after the end of the enrollment
  Analyze the number of patients treated with 3Dconformal Radiotherapy (3DCRT), Intensity Modulated Radiation Therapy (IMRT), Volumetric arch Therapy (VMAT), Tomotherapy, respectively with/without Image Guided Radiotherapy (IGRT) for pelvic irradiation
Outcome of treated prostate cancer | Three years after the end of the enrollment
  Biochemical relapse free survival
Outcome of treated prostate cancer | Three years after the end of the enrollment
  Clinical relapse free survival
Outcome of treated prostate cancer | Three years after the end of the enrollment
  Disease specific free survival
Outcome of treated prostate cancer | Three years after the end of the enrollment
  Overall survival
Toxicity of treated prostate cancer | Within 6 months after the end of the treatment
  register, using CTCAE v.4 acute and late urinary and rectal toxicities in the groups of patients treated with/without pelvic irradiation.
Comparison of toxicity and outcome in the different groups | Three years after the end of the enrollment
  Using chi-square test compare toxicities and clinical outcome in the different groups of patients.

CONTACTS AND LOCATIONS:
Overall Officials: Michela Buglione, Prof, Principal Investigator — University and Spedali Civili - Brescia
Locations (1):
- University and Spedali Civili - Brescia, Brescia, Italy

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-01-18): https://cdn.clinicaltrials.gov/large-docs/72/NCT03340272/Prot_SAP_000.pdf